CLINICAL TRIAL: NCT06561308
Title: A Single-arm, Multicenter Phase II Study of PD-1 Inhibitor Combined With Neoadjuvant Chemotherapy in Advanced Endometrial Cancer in Clinical Efficacy
Brief Title: Clinical Efficacy Study of PD-1 Inhibitor Combined With Neoadjuvant Chemotherapy in Advanced Endometrial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Xiangya Hospital of Central South University (Other); Tongji Hospital (Other); Qilu Hospital of Shandong University (Other); Anhui Provincial Cancer Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Henan Provincial People's Hospital (Other); Hunan Cancer Hospital (Other); Zhejiang Cancer Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Ningbo No. 1 Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO2024393
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-08

CONDITIONS: Endometrioid Endometrial Cancer
Keywords: Neoadjuvant chemotherapy; PD-1 inhibitor (Camrelizumab)
MeSH Terms: interventions — camrelizumab; Carboplatin; Paclitaxel; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Carboplatin AUC=4-6 q3w , paclitaxel 175 mg/m2 q3w and Camrelizumab iv.200mg q3w
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant chemotherapy combined with PD-1 inhibitor in FIGO III/IV Endometrial carcinoma (Experimental): Patients with advanced endometrial cancer were enrolled for 2-3 cycles of neoadjuvant chemotherapy in combination with camrelizumab, with imaging to assess efficacy; intermittent subtractive surgery (transabdominal hysterectomy + bilateral adnexectomies + pelvic lymph node dissection + pelvic and abdominal tumors resections +/- para-abdominal aortic lymph node dissection) was performed in patients with complete remissions (CR)/partial remissions (PR), and continued with 3-4 cycles of neoadjuvant chemotherapy in combination with camrelizumab.
  Interventions: Drug: Camrelizumab; Drug: Carboplatin; Drug: Paclitaxel; Procedure: Surgery

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab is administered at 200mg, q3w，intravenous infusion
Drug: Carboplatin — AUC=4-6，q3w，intravenous infusion
Drug: Paclitaxel — 175 mg/m2，q3w，intravenous infusion, administered over 30min.
Procedure: Surgery — Transabdominal hysterectomy + bilateral adnexectomy + pelvic lymph node dissection + pelvic-abdominal tumor resection +/- para-abdominal aortic lymph node dissection

SUMMARY:
Exploring the therapeutic effect of neoadjuvant chemotherapy combined with PD-1 inhibitor camrelizumab on advanced stage III-IV endometrial cancer

DETAILED DESCRIPTION:
Conduct domestic multicenter, prospective phase II single arm clinical trials to answer the following questions：

1. Evaluate the impact of neoadjuvant chemotherapy combined with camrelizumab on the remission rate, surgical complications, and surgical resection rate of advanced stage III-IV endometrial cancer;
2. Evaluate the effect of of neoadjuvant chemotherapy combined with camrelizumab on the survival of patients with advanced III-IV endometrial cancer;
3. Exploring the changes in tumor local immune related factors and cells before and after neoadjuvant chemotherapy and camrelizumab use, as well as the responsiveness of different molecular subtypes of endometrial cancer to neoadjuvant therapy, and screen for biological indicators that predict the effectiveness of camrelizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Endometrial cancer initially diagnosed as stage III non-operable resectable, stage IV (FIGO, 2009 criteria) after imaging evaluation
2. Pathologically confirmed endometrial cancer that looks like endometrial carcinoma
3. Patient age ≥18 years and ≤75 years old
4. ECOG status score of 0-1
5. tolerate surgery and radiotherapy
6. Laboratory tests: WBC ≥3.5×109/L, NEU ≥1.5×109/L, PLT ≥80×109/L, serum ≥80×109/L, serum ≥80×109/L, serum ≥80×109/L, serum ≥80×109/L.

   ×109/L, serum bilirubin ≤1.5 times the high limit of normal value, transaminase ≤1.5 times the high limit of normal value, BUN ≤1.5 times the high limit of normal value.

   1.5 times of the high limit of normal value, BUN, Cr≤normal value;
7. Able to follow up and good compliance;
8. Able to sign the informed consent form, including compliance with the requirements and restrictions listed in the informed consent form and the program.

Exclusion Criteria:

1. Subjects with an active, known, or suspected autoimmune disease, or a history of an autoimmune disease, except for: vitiligo, alopecia areata, Graves' disease, psoriasis, or eczema that has not required systemic therapy within the last 2 years, hypothyroidism that is asymptomatic or requires only stable doses of hormone replacement therapy (due to autoimmune thyroiditis), type 1 diabetes that requires only stable doses of insulin replacement therapy, asthma that subsides completely in childhood and does not require intervention in adulthood, or diseases that do not recur in the absence of external triggers;
2. Prior treatment with immune checkpoint inhibitors, including, but not limited to, other anti-PD-1, anti-PD-L1 antibodies, CTLA-4 antibodies, or any treatment directed against immune co-stimulators (e.g., antibodies directed against ICOS, CD40, CD137, GITR, OX40 targets, etc.) that target any mechanism of immune action against tumors;
3. Known hypersensitivity to any component and/or any excipient of the trial regimen;
4. Immunosuppressive drugs or systemic corticosteroids for immunosuppression (>10 mg/day of prednisone or other equivalent) within 2 weeks prior to trial dosing; topical, ophthalmic, intra-articular, intranasal, and inhaled corticosteroids are permitted;
5. Received herbs with antitumor effects or drugs with immunomodulatory effects (e.g., thymidine, interferon, interleukin-2) within 2 weeks prior to the trial;
6. Active systemic infection requiring systemic treatment;
7. Serious infection within 4 weeks prior to the first dose, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia;
8. Patients with untreated chronic hepatitis B, or HBV carriers with chronic hepatitis B virus (HBV) DNA greater than 1,000 IU/mL, or patients with active hepatitis C. Inactive HBsAg carriers, treated hepatitis B patients with stable disease (HBV DNA < 1000 IU/mL), and cured hepatitis C patients will be eligible for enrollment. HCV antibody-positive subjects will be eligible for the study only if they have a negative HCV RNA test;
9. Known active tuberculosis (TB), patients with suspected active TB should undergo chest X-ray and sputum examination in conjunction with clinical signs and symptoms for exclusion;
10. Immunodeficiency or human immunodeficiency virus (HIV antibody positive);
11. Subjects with active inflammatory bowel disease or a history of such disease (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea). Subjects who are unable to swallow or who have malabsorption syndrome, uncontrolled nausea, vomiting, diarrhea, or other gastrointestinal disorders that severely interfere with drug intake and absorption;
12. Known interstitial lung disease that is symptomatic or may interfere with detection or treatment of immune-associated pneumonia;
13. Treatment with a live or attenuated vaccine administered within 4 weeks prior to the first trial dose, inactivated seasonal influenza virus vaccine is permitted;
14. Patients who have received a prior allogeneic bone marrow transplant or solid organ transplant;
15. History of primary malignant tumor within the last 5 years;
16. Subjects who have undergone major surgery (e.g., open abdomen, open chest, organ resection, etc.) and severe trauma within 28 days prior to the first dose of implantable infusion devices are permitted;
17. Subjects with a history of gastrointestinal perforation, gastrointestinal fistula, or female genital fistula;
18. Uncontrolled other co-morbidities, symptoms, or medical history, including: (1) Persons with one of the following cardiovascular diseases or cardiovascular risk factors: myocardial infarction, unstable angina pectoris, pulmonary embolism, acute/continuous myocardial ischemia, cerebral vascular accident, transient ischemic attack, theor other clinically significant/required drug intervention arterial or venous thrombosis, embolism or cerebral ischemic events; symptoms of congestive heart failure (NYHA class III or higher) within 6 months (ii) clinically significant bleeding symptoms or a history of significant bleeding characteristics, such as gastrointestinal bleeding, gastric ulcer bleeding, or vasculitis, within 1 month prior to the first dose; (iii) clinically active hemoptysis, active diverticulitis, abdominal abscess, and gastrointestinal obstruction; (iv) uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage; (v) abnormalities of hepatic or renal development, or a history of surgery;
19. Female patients who are pregnant or breastfeeding; women of childbearing age who refuse to accept contraceptive measures during neoadjuvant immunotherapy;
20. Concurrent participation in other interventional clinical trials; participation in observational and non-interventional clinical trials is permitted;
21. Any condition that, in the opinion of the Investigator, may result in risk in the receipt of the study drug or that would interfere with the evaluation of the safety of the study drug or the interpretation of the study results. In the judgment of the Investigator, it is unlikely that Patients who, in the judgment of the Investigator, are less likely to comply with the study steps, restrictions, and requirements shall not be permitted to participate in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | At the end of the patient's treatment, up to 1 years.
  Proportion of patients with no tumor cells on postoperative pathology and negative lymph node metastasis

SECONDARY OUTCOMES:
Surgical complication rate | During and after the surgery, up to 2 years.
  intraoperative bleeding, vascular injuries, bladder injuries, rectal injuries, and ureteral injuries, as defined by the need for suture repair; occlusive nerve injuries, as defined by complete severance; and vascular injuries, as defined by the need to document the site of injury. Postoperative complications included: ureteral/bladder/rectal/vaginal fistula, internal hemorrhage, pelvic infection, lymphocyst, lymphatic fistula, lower extremity edema, lower extremity venous thrombosis, urinary retention, nerve injury, and bowel obstruction.
Adverse Event | during the treatment, up to 5 years.
  Adverse Effects of immunotherapy and chemotherapy
Remission rate (%) as assessed by RECIST 1.1 criteria | At the end of the patient's treatment, up to 1 years.
  Subjects were assessed for complete and partial remission rates according to RECIST 1.1 criteria
Event-free survival (EFS) | Until the end of the 3-year follow-up period, up to 5 years.
  the time between the enrollment and any documented tumor progression, recurrence, or death from any cause; the analysis of EFS includes the results of tumor evaluations during the study treatment and follow-up periods. If a patient had several indicators of PD or recurrence, the EFS analysis was performed using the indicator that appeared first; PD, recurrence, or death were considered to have reached the study endpoint; patients who were treated with other systemic or antitumor therapies directed at the target lesion of observation were also considered to be in PD; for patients who did not have PD, recurrence, or death at the end of the study, the time when the patient's failure to have a recurrence was last obtained was used as the time to censor the data.
Overall survival (OS) | Until the end of the 3-year follow-up period, up to 5 years.
  the time from the start of enrollment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wang, PHD, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's hospital school of medicine zhejiang university, Hangzhou, Zhejiang, China